CLINICAL TRIAL: NCT02387957
Title: A 24 Month Phase 2a Open Label, Randomized Study of Avastin®, Lucentis®, or Eylea® (Anti-VEGF Therapy) Administered in Combination With Fovista® (Anti-PDGF BB Pegylated Aptamer)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPH1006
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2019-02

CONDITIONS: Age-Related Macular Degeneration
Keywords: Wet AMD; subfoveal choroidal neovascularization; Fovista®; Avastin®; Lucentis®; Eylea®
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab; Ranibizumab; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fovista® plus bevacizumab (Experimental): Fovista® 1.5 mg intravitreal injection + bevacizumab 1.25 mg intravitreal injection
  Interventions: Drug: Fovista®; Drug: bevacizumab
- Fovista® plus ranibizumab (Experimental): Fovista® 1.5 mg intravitreal injection + 0.5 mg ranibizumab intravitreal injection
  Interventions: Drug: Fovista®; Drug: ranibizumab
- Fovista® plus aflibercept (Experimental): Fovista® 1.5 mg intravitreal injection + 2.0 mg aflibercept intravitreal injection
  Interventions: Drug: Fovista®; Drug: aflibercept

INTERVENTIONS:
Drug: Fovista®
Drug: bevacizumab
  Other Names: Avastin®
  Arms: Fovista® plus bevacizumab
Drug: ranibizumab
  Other Names: Lucentis®
  Arms: Fovista® plus ranibizumab
Drug: aflibercept
  Other Names: Eylea®
  Arms: Fovista® plus aflibercept

SUMMARY:
To evaluate the safety of intravitreal (IVT) Fovista® administered in combination with anti-VEGF therapy.

DETAILED DESCRIPTION:
60 subjects randomized 1:1:1 and treated with IVT Fovista® 1.5 mg/eye in combination with anti-VEGF therapy as follows:

* Avastin® 1.25 mg/eye (20 subjects)
* Lucentis® 0.5 mg/eye (20 subjects)
* Eylea® 2.0 mg/eye (20 subjects)

Subjects will be stratified by lesion size (≤2 DA vs. >2 DA).

Subjects will be treated with "combination therapy" of IVT Fovista® and IVT anti-VEGF therapy every month for the first 5 months (Day 1, Months 1,2,3,4), followed by Q12W (every 12 weeks) administration (Months 7,10, 13,16, 19 and 22), for a total of 24 months.

When administered, IVT Fovista® will be given first, followed by IVT anti-VEGF (same day).

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender aged ≥ 50 years.
* Active subfoveal choroidal neovascularization (CNV) due to AMD.

Exclusion Criteria:

* Any intraocular surgery or thermal laser within three (3) months of trial entry. Any prior thermal laser in the macular region, regardless of indication.
* Subjects with subfoveal scar or subfoveal atrophy
* Any ocular or periocular infection in the past twelve (12) weeks.
* History of any of the following conditions or procedures in the study eye: Rhegmatogenous retinal detachment, pars plana vitrectomy, filtering surgery (e.g. trabeculectomy), glaucoma drainage device, corneal transplant.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Phoenix, Arizona
  - Beverly Hills, California
  - Sacramento, California
  - Santa Ana, California
  - New London, Connecticut
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Augusta, Georgia
  - Oak Forest, Illinois
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Reno, Nevada
  - Rochester, New York
  - Cleveland, Ohio
  - Huntingdon Valley, Pennsylvania
  - Ladson, South Carolina
  - Abilene, Texas
  - Amarillo, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Silverdale, Washington
  - Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

RESULTS

PARTICIPANT FLOW:
Groups:
- Fovista® Plus Bevacizumab: Fovista® 1.5 mg intravitreal injection + bevacizumab 1.25 mg intravitreal injection
  Fovista®
  bevacizumab
- Fovista® Plus Ranibizumab: Fovista® 1.5 mg intravitreal injection + 0.5 mg ranibizumab intravitreal injection
  Fovista®
  ranibizumab
- Fovista® Plus Aflibercept: Fovista® 1.5 mg intravitreal injection + 2.0 mg aflibercept intravitreal injection
  Fovista®
  aflibercept
Period: Overall Study
Arm/Group | Fovista® Plus Bevacizumab | Fovista® Plus Ranibizumab | Fovista® Plus Aflibercept
Started | 21 | 21 | 21
Completed | 0 (The study was discontinued) | 0 (The study was discontinued) | 1 (The study was discontinued)
Not Completed | 21 | 21 | 20
Not completed — The study was discontinued | 21 | 21 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fovista® Plus Bevacizumab | Fovista® Plus Ranibizumab | Fovista® Plus Aflibercept | Total
Number analyzed (Participants) | 21 | 21 | 21 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 8
  >=65 years | 18 | 18 | 19 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.5 (9.51) | 77.2 (10.43) | 77.9 (8.99) | 77.9 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 15 | 44
  Male | 8 | 5 | 6 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 21 | 21 | 20 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 21 | 63

OUTCOME MEASURES:

1. Primary Outcome: Total Numer of Systemic Adverse Events
Description: Number of Patients with Systemic Adverse Events
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Fovista® Plus Bevacizumab | Fovista® Plus Ranibizumab | Fovista® Plus Aflibercept
Number analyzed (Participants) | 21 | 21 | 21
Participants | 3 | 3 | 5

2. Primary Outcome: Total Number of Other Adverse Events (>5%)
Description: Number of Patients with Other Adverse Events
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Fovista® Plus Bevacizumab | Fovista® Plus Ranibizumab | Fovista® Plus Aflibercept
Number analyzed (Participants) | 21 | 21 | 21
Participants | 15 | 16 | 16

ADVERSE EVENTS:
Time Frame: Up to a maximum exposure of 24 months
Arm/Group | Fovista® Plus Bevacizumab | Fovista® Plus Ranibizumab | Fovista® Plus Aflibercept
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/21 | 3/21 | 5/21
Other Adverse Events (participants affected / at risk) | 15/21 | 16/21 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fovista® Plus Bevacizumab (N=21) | Fovista® Plus Ranibizumab (N=21) | Fovista® Plus Aflibercept (N=21)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cervical spine stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified reccurent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fovista® Plus Bevacizumab (N=21) | Fovista® Plus Ranibizumab (N=21) | Fovista® Plus Aflibercept (N=21)
Neovascular age-related macular degeneration (Eye disorders) | 4 (4) | 1 (1) | 6 (6)
Cataract (Eye disorders) | 1 (1) | 3 (6) | 4 (4)
Eye pain (Eye disorders) | 4 (4) | 0 (0) | 4 (6)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 4 (5)
Vitreous floaters (Eye disorders) | 1 (1) | 2 (2) | 3 (3)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Conjuctival haemorrhage (Eye disorders) | 7 (11) | 6 (16) | 1 (1)
Eye irritation (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1) | 3 (3) | 1 (1)
Vitreous detachment (Eye disorders) | 2 (2) | 2 (2) | 0 (0)
Seasonal allergy (General disorders) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (5) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Intraocular pressure increased (Investigations) | 3 (6) | 2 (4) | 6 (9)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Ocular Discomfort (Eye disorders) | 2 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution agrees not to individually publish the results of the Study without Ophthotech's prior written consent. Institution may participate in a joint, multi-center publication of the Study results with other investigators and/or institutions only, upon the prior written consent of Ophthotech.